CLINICAL TRIAL: NCT06911203
Title: A Phase II, Randomized Open-label, Multicenter Study to Evaluate the Efficacy and Safety of BGM0504 Compared to Tirzepatide in Adults Who Have Obesity
Brief Title: A Study of BGM0504 in Participants With Obesity
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: BrightGene Bio-Medical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BGM0504-II -WL-02
Record Dates: First submitted 2025-04-03; First posted 2025-04-04 (Actual); Last update posted 2025-10-28 (Actual); Status verified 2025-01

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Tirzepatide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- BGM0504 (Experimental): Participants will receive BGM0504 subcutaneously(SC).
  Interventions: Drug: BGM0504
- Tirzepatide (Active Comparator): Paritcipants will receive tirzepatide SC.
  Interventions: Drug: Tirzepatide

INTERVENTIONS:
Drug: BGM0504 — Administered SC
  Arms: BGM0504
Drug: Tirzepatide — Administered SC
  Arms: Tirzepatide

SUMMARY:
To evaluate the efficacy and safety of BGM0504 compared with Tirzepatide in adult participants who have obesity without diabetes after 26 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

* ● Able and willing to provide a written informed consent.

  * Male or female subjects, 18-65 years of age at the time of signing informed consent.
  * At screening visit, 35.0 ﹤BMI﹤ 45.0 kg/m2;
  * Diet and exercise control for at least 3 months before screening visit, and be of stable weight (± 5%) self-reported change within the last 3 months.

Exclusion Criteria:

* ●History of chronic or acute pancreatitis.

  * History of severe drug allergy or specific allergic disease or severe allergies.
  * Family or personal history of medullary thyroid carcinoma (MTC) or multiple endocrine neoplasia syndrome type 2(MEN-2).
  * History of malignant tumors [except carcinoma in situ with no recurrence within 5 years (except for malignant melanoma in situ), skin basal cell carcinoma and squamous cell carcinoma].
  * Suspected or confirmed history of alcohol or drug abuse;
  * Any chronic infections likely to interfere with study conduct or interpretation such as hepatitis B (HBV), hepatitis C (HCV), human immunodeficiency virus (HIV) or treponema pallidum (TP).
  * Donation or loss of 400 mL or more of blood within 3 months prior to screening, or blood donation during screening or within 3 months after the end of the trial.
  * Pregnant or lactating woman.
  * Any disorder, unwillingness, or inability not covered by any of the other exclusion criteria, which in the Investigator's opinion, might jeopardize the participant's safety or compliance with the protocol.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-04-03 (Actual); Primary Completion 2026-01-11 (Estimated); Study Completion 2026-01-11 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline in Body Weight | Week 0, Week 26
  Change from baseline in body weight after 26 weeks of treatment

SECONDARY OUTCOMES:
Change From Baseline in BMI | Week 18, Week 26
  Change from baseline in BMI after 26 weeks of treatment
Change From Baseline in Waist Circumference | Week 18, Week 26
  Change from baseline in waist circumference after 26 weeks of treatment
Change from Baseline in Systolic Blood Pressure (SBP) | Week 18, Week 26
  Change from Baseline in SBP after 26 weeks of treatment
Change from Baseline in Diastolic Blood Pressure (DBP) | Week 18, Week 26
  Change from Baseline in DBP after 26 weeks of treatment
Change from Baseline in Impact of Weight on Quality of Life-Lite Clinical Trials Version (IWQOL-Lite-CT) | Week 0, Week 26
  Change from Baseline in IWQOL-Lite-CT after 26 weeks of treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China